CLINICAL TRIAL: NCT02877836
Title: Functional Magnetic Resonance and Diffusion Tensor Imaging in the Preoperative Assessment of Dystonia
Brief Title: Functional MRI and DTI in the Preoperative Assessment of Dystonia
Acronym: IRMF-DIFF
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: end of inclusion period and difficulties on recruitment of one patient group
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 9095
Record Dates: First submitted 2016-07-06; First posted 2016-08-24 (Estimated); Last update posted 2021-12-28 (Actual); Status verified 2021-12

CONDITIONS: Isolated Cervical Dystonia; Complex Dystonia; Spasticity
Keywords: Dystonia; fMRI; DTI; DBS
MeSH Terms: conditions — Muscle Spasticity; Dystonia | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Segmentary dystonia (Other): to identify movement-related functional magnetic resonance imaging (fMRI) activation patterns
  Interventions: Other: magnetic resonance imaging (fMRI)
- Hemidystonia (Other): to identify movement-related functional magnetic resonance imaging (fMRI) activation patterns
  Interventions: Other: magnetic resonance imaging (fMRI)
- Generalized dystonia (Other): to identify movement-related functional magnetic resonance imaging (fMRI) activation patterns
  Interventions: Other: magnetic resonance imaging (fMRI)
- Healthy control subjects (Other): to identify movement-related functional magnetic resonance imaging (fMRI) activation patterns
  Interventions: Other: magnetic resonance imaging (fMRI)

INTERVENTIONS:
Other: magnetic resonance imaging (fMRI) — To identify movement-related fMRI activation pattern in dystonic patients in comparison to healthy controls Assessment of white matter integrity in the corticospinal tract in a group og dystonic patients compared with the healthy control group

SUMMARY:
The aim of this study is to evaluate the organization of the motor circuit in a group of patients suffering from dystonia compared with a group of healthy controls. Deep Brain stimulation is a functional neurosurgery technique consisting in neuromodulation of the motor circuit that has been applied to dystonia. The efficiency of this technique depends on the relative preservation of the function and the structure of the motor network .

The assessment of neuronal circuit by advanced techniques of functional neuroimaging in this study might contribute to expand our understanding of the abnormalities in motor circuit activation and the integrity of CNS structure underlying dystonia. This study might contribute therefore to the refinement of Deep brain stimulation indications and techniques in complex dystonia syndromes

DETAILED DESCRIPTION:
Advances in the field of functional neurosurgery, neuroradiology and virus neuronal tracing studies have expanded our knowledge of the circuits underlying the clinical expression of several neurologic syndromes. Globus pallidus internus (GPi) Deep brain stimulation (DBS) is a validated technique for the treatment of 'isolated dystonia'. The efficiency of this therapy in 'complex dystonia', commonly associated with focal brain lesions, is limited and heterogeneous. Broadening indications for DBS therapy to complex DDS disorders require further improvement of preoperative assessment of motor circuit functional reorganization and white matter integrity. The efficacy of neuromodulation in these clinical syndromes is determined by the severity of pyramidal involvement, the interactions between cortico-striato-pallido-thalamic and cerebello-thalamo-cortical circuits and motor network reorganization at the cortical level.

The aim of the study is to identify movement-related functional magnetic resonance imaging (fMRI) activation patterns in a group of dystonic patients in comparison to healthy controls (HC). Further analysis will assess the recruitment pattern in different patient subgroups defined according to clinical and radiological criteria relevant to GPi DBS eligibility (hyperkinetic/ hypokinetic and prepallidal/ postpallidal). Diffusion tensor imaging (DTI) will be applied to the assessment of the topographic distribution and severity of white matter lesions in the group of dystonic patients in comparison with HC.

Further knowledge concerning motor network organization and white matter integrity after focal brain lesions might contribute to the understanding of this mitigated response to DBS and to the refinement of DBS indications and techniques in secondary dystonia

ELIGIBILITY:
Inclusion Criteria:

* Age limits ≥ 18 et < 85 years
* Right-handed patients/healthy controls, according to Edinburgh Handedness Inventory
* The participating subjects must be affiliated to the French public health system
* Written consent to participate in this study

For the patients

* Patients affected by isolated or complex dystonia admitted to hospital in the Unit of Functional Neurosurgery in order to assess eligibility for deep cerebral stimulation therapy
* Ability to understand the instructions to perform the experimental paradigm (the motor task) used in the design of the functional MRI

For the healthy control subjects :

* Absence of current neurologic pathology
* Absence of personal history of neurologic pathology, including perinatal anoxic injury, meningitis, vascular, metabolic, inflammatory pathology, epilepsy, cranial trauma with loss of consciousness or with associated neurological symptoms.
* Absence of orthopaedic injury in the upper limbs

Exclusion Criteria:

* Non Specific criteria

  * Contraindication for the realization of a MRI (pacemaker, valve prothesis non compatible with MRI, cochlear implant, aneuvrysmal clip, presence of an Intra-ocular metallic foreign object or coronary endoprosthesis)
  * Pregnancy, breastfeeding
  * Adults protected by the law
* Non Specific criteria • Severe dyskinesia preventing the realization of motor task during functional MRI without general anesthesia

Ages: 18 Years to 84 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2014-09-19 (Actual); Primary Completion 2016-06-03 (Actual); Study Completion 2016-06-03 (Actual)

PRIMARY OUTCOMES:
Integrity of Motor circuit reorganization in dystonia | 1 day
  All the subjects participating in the study will undergo a Functional MRI study with a 'box and block' design comparing brain activity during the execution of a motor task and rest. Resting state fMRI will also be recorded. Statistical Parametric Mapping (SPM8) software will be used in order to perform spatially extended statistical processes to test the hypothesis whether there is a difference between both groups in functional imaging data. This analysis will provide a statistical map showing the clusters of brain activation where there is a significant difference between the group of dystonic patients and the group of healthy controls
Integrity of corticospinal tract white matter in dystonia | 1 day
  Fractional anisotropy (FA) is a measure derived of Diffusion tensor imaging that quantifies the degree of directionality of the local tract structure. This parameter is considered to be a marker for white matter tract integrity.
  FSL software will be used to analyse Diffusion Tensor Imaging (DTI) data
  1. Tract-based spatial statistics (TBSS) will be used to obtain a voxelwise statistical map comparing fractional anisotropy in the major tracts in the group ot dystonic patients and the group of healthy controls.
  2. Probabilistic tractography will be used to obtain tract-derived DTI parameters in the corticospinal and thalamocortical tracts that will be correlated with clinical scales (Burke-Fahn-Marsden Dystonia scale). Several DTI parameters will be analysed: mean fractional anisotropy, mean diffusivity, parallel and perpendicular diffusivity

SECONDARY OUTCOMES:
Movement-related fMRI activation pattern in dystonic patients | 1 day
  To identify movement-related fMRI activation pattern in different subgroups of dystonic patients classified following clinical (hyperkinetic versus hypokinetic) and radiologic criteria (prepallidal versus postpallidal lesions) Statistical Parametric Mapping (SPM8) software will be used to test the hypothesis whether patients with different clinical phenotypes (hyperkinetic versus hypokinetic) or patients with different radiologic presentation (prepallidal versus postpallidal lesions) show significant differences in the pattern of brain activation related to the execution of a motor task.
  This analysis will provide a statistical map showing the clusters of brain activation where there is a significant difference between both groups

CONTACTS AND LOCATIONS:
Overall Officials: Victoria Gonzalez, MD PhD, Principal Investigator — CHU de Montpellier
Locations (1):
- CHU de Montpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: No